CLINICAL TRIAL: NCT06567873
Title: Assessment of Preoperative Gastric Content With Ultrasound in Patients Reporting Cannabis Use
Brief Title: Gastric Ultrasound Assessment for Patients Taking Cannabis
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1155
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Gastric Ultrasound; Point of Care Ultrasound; Cannabis Use
Keywords: cannabis; gastric ultrasound
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cannabis Users: The cannabis user group will be comprised of patients who report preoperative cannabis use within 1 month of surgery date. This group will receive the ultrasound exam to assess stomach contents.
  Interventions: Other: Gastric Ultrasound Exam

INTERVENTIONS:
Other: Gastric Ultrasound Exam — A gastric ultrasound is a simple, fast, non-invasive bedside diagnostic test that provides a qualitative and quantitative assessment of gastric contents. There are no known risks of a gastric ultrasound exam.

SUMMARY:
The aim of this study is to perform bedside gastric point of care ultrasound (POCUS) exams to assess the gastric volume and content (clear liquids vs solid food) perioperatively in patients who report cannabis use.

DETAILED DESCRIPTION:
Cannabis use in the United States has continued to increase in recent years, particularly in the adult population. Ease of access through legalization paired with improved public perception has contributed to the uptick in cannabis use. The subset of cannabis users suffering from pain who present for surgery pose a risk for perioperative aspiration due to the slowing of gastric motility due to cannabis use. There is currently no adapted NPO guideline to account for cannabis use.

Gastric Ultrasound (GUS) can be used as a bedside tool for assessing a patient's stomach contents and risk of aspiration. GUS can identify whether a patient's stomach is empty or filled with clear liquid, thick liquid, or solid food. The volume of the stomach can be accurately calculated if there is clear liquid content. A full stomach is categorized as those with solid or thick liquid content or with clear liquid measuring more than 1.5 ml/kg body weight. As GUS is noninvasive and does not pose risk to patients, it is a useful tool assessing aspiration risk in the preoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Any patient reporting preoperative cannabis usage within 1 month of surgery date

Exclusion Criteria:

* Patient refusal to participate
* Patient with gastric bypass or any other gastric surgery
* Large hiatal hernia
* Patients with large ascites
* Patients on peritoneal dialysis
* Emergency surgery
* Pre-existing diagnosis of gastroparesis
* Parkinson's disease
* Diabetes
* Currently taking metformin
* Chronic kidney disease stage 3 or higher
* Creatinine ≥ 1.2
* Esophageal surgery
* Currently taking GLP1 agonist medication

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of patients scheduled for surgery at HSS who meet the following inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Incidence of delayed gastric emptying | This will be measured pre-operatively in the holding room area.
  A full stomach on gastric ultrasound is defined by the presence of either solid food, thick liquids, or a specific volume (>1.5 ml/kg) of clear liquids on gastric ultrasound.

SECONDARY OUTCOMES:
Nothing by mouth (NPO) intervals | This will be measured pre-operatively in the holding room area.
  Measure the NPO interval after last solid food and liquid consumption
Presence of gastric peristalsis | This will be measured pre-operatively in the holding room area.
  Gastric peristalsis will be graded as absent, slow, or normal on gastric ultrasound
Time interval since last cannabis use | This will be measured pre-operatively in the holding room area.
  Measure the time from last cannabis consumption to the time the gastric ultrasound was performed

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Panzer, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King DD, Stewart SA, Collins-Yoder A, Fleckner T, Price LL. Anesthesia for Patients Who Self-Report Cannabis (Marijuana) Use Before Esophagogastroduodenoscopy: A Retrospective Review. AANA J. 2021 Jun;89(3):205-212. PMID 34042571
- [Background] Cammarano CA, Villaluz JE. A Reason to Rethink Fasting Guidelines? Marijuana-Induced Gastroparesis and the Implications for Aspiration Risk in the Nil Per Os (NPO) Patient: A Case Report. Am J Case Rep. 2021 Nov 29;22:e934187. doi: 10.12659/AJCR.934187. PMID 34840324
- [Background] McCallum RW, Soykan I, Sridhar KR, Ricci DA, Lange RC, Plankey MW. Delta-9-tetrahydrocannabinol delays the gastric emptying of solid food in humans: a double-blind, randomized study. Aliment Pharmacol Ther. 1999 Jan;13(1):77-80. doi: 10.1046/j.1365-2036.1999.00441.x. PMID 9892882
- [Background] Esfandyari T, Camilleri M, Ferber I, Burton D, Baxter K, Zinsmeister AR. Effect of a cannabinoid agonist on gastrointestinal transit and postprandial satiation in healthy human subjects: a randomized, placebo-controlled study. Neurogastroenterol Motil. 2006 Sep;18(9):831-8. doi: 10.1111/j.1365-2982.2006.00834.x. PMID 16918762